CLINICAL TRIAL: NCT05163327
Title: Oxygen-enhanced Magnetic Resonance Imaging (OE-MRI) of the Heart: A Feasibility Study
Acronym: OE-MRI
Status: Withdrawn | Type: Observational
Why Stopped: Accumulated evidence (including data acquired in parallel studies, in other centres and in published literature) suggest that the technique was unlikely to produce a signal in the heart.
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: Cardiac-OE-MRI-01
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease
Keywords: MRI, Imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: 10 Volunteers (Male or Female), aged18 or over, with no known history of Coronary Artery Disease
  Interventions: Procedure: Oxygen-enhanced Cardiac MRI
- Known Coronary Artery Disease: 10 Volunteers (Male orFemale), aged 18 or over,with a known significant (defined as => 70% stenosis) single or 2 vessel Coronary Artery Disease
  Interventions: Procedure: Oxygen-enhanced Cardiac MRI

INTERVENTIONS:
Procedure: Oxygen-enhanced Cardiac MRI — The MRI scan will include assessment of cardiac function. Myocardial magnetic properties (T1, T2, T2*) will be measured while patients are breathing room air, oxygen and during an infusion of adenosine. The scan will last for approximately 60 minutes. Prior to the scan patients will have an intravenous cannula (venflon) placed in an arm vein.

SUMMARY:
This exploratory pilot study aims to set up cardiac oxygen enhanced magnetic resonance imaging (OE-MRI). It will involve 10 healthy volunteers and 10 patients with known coronary artery disease (CAD) having a MRI scan.

If positive, this data would be used to power an appropriately sized study assessing the utility of cardiac OE-MRI in CAD and other cardiac pathologies.

DETAILED DESCRIPTION:
Determining the presence and severity of myocardial ischaemia is a key goal in the effective management of coronary artery disease (CAD). Untreated ischaemia is an important determinant of adverse outcome, and the benefits of ischemia-driven revascularization are well recognized.1

Anatomic appearances of coronary artery disease are poorly predictive of myocardial ischemia.1 2 Therefore, concurrent assessment of the functional severity of coronary stenosis is used to guide revascularization.3 In the clinical setting, a number of imaging methods are available, including nuclear techniques, echocardiography, and cardiovascular magnetic resonance (CMR). Such modalities assess flow heterogeneity and contractile abnormalities, but these serve as surrogates of myocardial ischemia: ischemia per se is not measured. Furthermore, these functional imaging modalities rely on the use of exogenous contrast agents, which, albeit small, carry additional risks and can be contraindicated in certain populations.

Blood oxygen level dependent (BOLD) imaging exploits the inherent paramagnetic properties of haemoglobin.4 The transition from diamagnetic oxyhaemoglobin to paramagnetic deoxyhaemoglobin induces magnetic susceptibility differences, resulting in a change in magnetic resonance signal intensity and thereby generating oxygen dependent contrast. Thus BOLD imaging provides insight into myocardial tissue oxygenation. Since hypoxia is the initiator of the ischaemic cascade, assessment of regional myocardial oxygenation with BOLD imaging has been hypothesised to reflect more directly the imbalance between oxygen supply and demand and be sensitive for detecting CAD. Indeed initial evaluation of BOLD imaging for detecting CAD has produced promising results.5-7 Furthermore, BOLD has provided pathological insight into other myocardial pathologies. Myocardial perfusion (blood flow) can be dissociated from oxygenation i.e. hypoperfusion is not necessarily commensurate with tissue hypoxia. For example, myocardial oxygen demand may be down-regulated in hibernating myocardium, and may be upregulated in hypertrophic cardiomyopathy (HCM) due to the increased cost of energy metabolism. In HCM mutation carriers without left ventricular hypertrophy, Karamitsos et al demonstrated normal myocardial perfusion reserve, but abnormal myocardial oxygenation during stress, possibly explained by the fact that sarcomere gene mutations increase the energy cost of contraction before the onset of hypertrophy.8

However, BOLD imaging is associated with a number of disadvantages. First, since the BOLD signal reflects deoxyhaemoglobin which is confined to blood vessels, it doesn't truly reflect tissue oxygen status.9 Second, the BOLD signal is also dependent on vessel geometry, changes in blood flow and blood volume, which thus can confound the signal.9 Finally, the CMR techniques used to measure the BOLD signal (T2* of T2) are not quantitative since a change in T2* or T2 cannot be related to a change in the partial pressure of oxygen (PO2). Instead, semi-quantitative measurements are made using signal intensity and are assumed to reflect oxygenation.

Oxygen enhanced magnetic resonance imaging (OE-MRI) potentially overcomes these limitations. Oxygen itself has paramagnetic properties; it increases the proton longitudinal relaxation rate (R1) of water containing dissolved oxygen.10 The measured change in R1 (= 1/T1, where T1 relaxation time is an inherent magnetic property of all tissues) induced by breathing oxygen is directly proportional to the change in PO2. In OE-MRI the change in R1 on breathing elevated concentrations of oxygen is measured. The benefits of OE-MRI over BOLD are therefore that it is sensitive to tissue oxygenation, it is not dependent on changes in blood flow and volume, and it is truly quantitative, since the change in R1 is directly proportional to the change in PO2. Thus it potentially offers a quantitative measure of myocardial oxygenation. OE-MRI has been used to assess lung tissue oxygenation,11 solid tumour oxygenation12 and to assess placental oxygenation in pregnant women13 on conventional clinical MRI scanners with very encouraging results.

OE-MRI has not been applied in the heart. We hypothesise that OE-MRI will allow non-invasive, non-ionising, and quantitative assessment of myocardial tissue oxygenation, that is free from exogenous contrast agent. If this is the case, OE-MRI will offer enormous potential in terms of the diagnosis and management of CAD, and in terms of providing pathophysiological insight into cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* 10 healthy volunteers and 10 patients with known significant (defined as > 70% stenosis) single or 2 vessel CAD
* Male or female > 18 years of age
* Females will be non-pregnant and non-lactating

Exclusion Criteria:

* Contraindication to MRI (including claustrophobia)
* History of any significant lung disease including asthma and COPD
* History of type II respiratory failure
* Second degree and higher atrio-ventricular conduction delay
* Patients taking Dipyridamole, or theophylline-based medication
* Significant left main stem coronary artery disease
* Recent myocardial infarction (within 2 months)
* Unstable angina
* Abnormal heart rhythm e.g. atrial fibrillation, atrial flutter, atrial or ventricular bigeminy
* Pregnancy/breast-feeding. Women of childbearing potential (not >2 years post- menopausal and/or not surgically sterilised) must have a negative blood serum pregnancy test.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ten healthy volunteers and 10 patients with CAD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To apply OE-MRI in the heart and compare it to BOLD imaging | 24 Months
  To apply OE-MRI in the heart and compare it to BOLD imaging

CONTACTS AND LOCATIONS:
Overall Officials: Chris Miller, MBChB, MRCP, Principal Investigator — Manchester University NHS FT
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Uren NG, Melin JA, De Bruyne B, Wijns W, Baudhuin T, Camici PG. Relation between myocardial blood flow and the severity of coronary-artery stenosis. N Engl J Med. 1994 Jun 23;330(25):1782-8. doi: 10.1056/NEJM199406233302503. PMID 8190154
- [Background] Kern MJ, Lerman A, Bech JW, De Bruyne B, Eeckhout E, Fearon WF, Higano ST, Lim MJ, Meuwissen M, Piek JJ, Pijls NH, Siebes M, Spaan JA; American Heart Association Committee on Diagnostic and Interventional Cardiac Catheterization, Council on Clinical Cardiology. Physiological assessment of coronary artery disease in the cardiac catheterization laboratory: a scientific statement from the American Heart Association Committee on Diagnostic and Interventional Cardiac Catheterization, Council on Clinical Cardiology. Circulation. 2006 Sep 19;114(12):1321-41. doi: 10.1161/CIRCULATIONAHA.106.177276. Epub 2006 Aug 28. PMID 16940193
- [Background] Pauling L, Coryell CD. The Magnetic Properties and Structure of Hemoglobin, Oxyhemoglobin and Carbonmonoxyhemoglobin. Proc Natl Acad Sci U S A. 1936 Apr;22(4):210-6. doi: 10.1073/pnas.22.4.210. No abstract available. PMID 16577697
- [Background] Arnold JR, Karamitsos TD, Bhamra-Ariza P, Francis JM, Searle N, Robson MD, Howells RK, Choudhury RP, Rimoldi OE, Camici PG, Banning AP, Neubauer S, Jerosch-Herold M, Selvanayagam JB. Myocardial oxygenation in coronary artery disease: insights from blood oxygen level-dependent magnetic resonance imaging at 3 tesla. J Am Coll Cardiol. 2012 May 29;59(22):1954-64. doi: 10.1016/j.jacc.2012.01.055. PMID 22624835
- [Background] Karamitsos TD, Leccisotti L, Arnold JR, Recio-Mayoral A, Bhamra-Ariza P, Howells RK, Searle N, Robson MD, Rimoldi OE, Camici PG, Neubauer S, Selvanayagam JB. Relationship between regional myocardial oxygenation and perfusion in patients with coronary artery disease: insights from cardiovascular magnetic resonance and positron emission tomography. Circ Cardiovasc Imaging. 2010 Jan;3(1):32-40. doi: 10.1161/CIRCIMAGING.109.860148. Epub 2009 Nov 17. PMID 19920032
- [Background] Friedrich MG, Niendorf T, Schulz-Menger J, Gross CM, Dietz R. Blood oxygen level-dependent magnetic resonance imaging in patients with stress-induced angina. Circulation. 2003 Nov 4;108(18):2219-23. doi: 10.1161/01.CIR.0000095271.08248.EA. Epub 2003 Oct 13. PMID 14557359
- [Background] Karamitsos TD, Dass S, Suttie J, Sever E, Birks J, Holloway CJ, Robson MD, Jerosch-Herold M, Watkins H, Neubauer S. Blunted myocardial oxygenation response during vasodilator stress in patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2013 Mar 19;61(11):1169-76. doi: 10.1016/j.jacc.2012.12.024. PMID 23498131
- [Background] Padhani AR, Krohn KA, Lewis JS, Alber M. Imaging oxygenation of human tumours. Eur Radiol. 2007 Apr;17(4):861-72. doi: 10.1007/s00330-006-0431-y. Epub 2006 Oct 17. PMID 17043737
- [Background] Young IR, Clarke GJ, Bailes DR, Pennock JM, Doyle FH, Bydder GM. Enhancement of relaxation rate with paramagnetic contrast agents in NMR imaging. J Comput Tomogr. 1981 Dec;5(6):543-7. doi: 10.1016/0149-936x(81)90089-8. PMID 7053127
- [Background] Kershaw LE, Naish JH, McGrath DM, Waterton JC, Parker GJ. Measurement of arterial plasma oxygenation in dynamic oxygen-enhanced MRI. Magn Reson Med. 2010 Dec;64(6):1838-42. doi: 10.1002/mrm.22571. PMID 20677232
- [Background] O'Connor JP, Naish JH, Parker GJ, Waterton JC, Watson Y, Jayson GC, Buonaccorsi GA, Cheung S, Buckley DL, McGrath DM, West CM, Davidson SE, Roberts C, Mills SJ, Mitchell CL, Hope L, Ton NC, Jackson A. Preliminary study of oxygen-enhanced longitudinal relaxation in MRI: a potential novel biomarker of oxygenation changes in solid tumors. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1209-15. doi: 10.1016/j.ijrobp.2008.12.040. Epub 2009 Mar 26. PMID 19327904
- [Background] Huen I, Morris DM, Wright C, Parker GJ, Sibley CP, Johnstone ED, Naish JH. R1 and R2 * changes in the human placenta in response to maternal oxygen challenge. Magn Reson Med. 2013 Nov;70(5):1427-33. doi: 10.1002/mrm.24581. Epub 2012 Dec 27. PMID 23280967